CLINICAL TRIAL: NCT04381585
Title: Efficacy of Distraction Osteogenesis in Vertically Deficient Anterior Maxillary and Mandibular Bone by Using Mini Distractor With a Submerged Activation Component. A Clinical and Radiographical Study
Brief Title: Mini Distractor in Vertically Deficient Bone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SVS Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, Dr R Viswa Chandra, Primary Investigator, SVS Institute of Dental Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SVSIDS/PERIO/4/2019
Record Dates: First submitted 2020-04-29; First posted 2020-05-11 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Periodontitis; Alveolar Bone Loss
MeSH Terms: conditions — Periodontitis; Alveolar Bone Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Distraction osteogenesis using mini distractor (Experimental): A mini distractor will be used to move bone. Distraction osteogenesis originally developed for the severe craniofacial malformations has been adapted to correct vertical defects of the oral bone to improve bone volume for dental procedures.
  However, the design of the distractor
  1. has not evolved to adapt to a much smaller surgical site such as bone ridge in the oral cavity which necessitates a smaller screw.
  2. are bulky, cumbersome to place, and cause significant discomfort to the patient.
  3. has an extraoral component jutting out of the mouth to which a key (blue object) is attached to turn the screw to move bone fragments. Our Solution and the Innovation is to remove the extra-oral component by reducing the size and permitting an atraumatic placement of the screw under the gingiva (gum) thereby lessening irritation for the patient.
  Interventions: Device: A MINI DISTRACTOR WITH A SUBMERGED ACTIVATION COMPONENT

INTERVENTIONS:
Device: A MINI DISTRACTOR WITH A SUBMERGED ACTIVATION COMPONENT — Mini distractor is used to regenerate alveolar bone which is resorbed due various reasons. The distractor uses a winch-like submucosal activation component which is buried in the tissue; Flicking the winch turns the screw which moves the segment upwards in the direction of black arrow increasing height.

SUMMARY:
ADO is a bone regeneration technique, introduced by Chin and Toth in 1996 based in a biological process used for regenerate and consolidate bone between two bone segments obtained after osteotomy.These segments have been gradually separated by the process of distraction. ADO can be performed both horizontally (AHDO) and vertically (AVDO).

DETAILED DESCRIPTION:
Distraction osteogenesis (DO) can be used to regenerate missing hard and soft tissue, Distraction osteogenesis relies on the body's ability to generate bone as two segments of bone are "distracted" apart. The osteotomies are created and the distraction device is placed. Typically, there is a latency phase of one week were a ﬁbrovascular bridge is formed in the osteotomy site. This provides a template to generate new bone as the segments are distracted apart during the activation phase. Once the desired distraction has occurred, the device is left in place for a period of time. Once consolidation (typically 2 to 6 months) has occurred, the distraction device can be removed and implants can be placed. Chiapasco compared GBR to DO and found that both are equally effective in alveolar bone augmentation for implant placement and further stated that the long-term prognosis of vertical bone gain in DO is more predictable.

ELIGIBILITY:
Inclusion Criteria:

* Acquired alveolar defects (Post extraction, Traumatic avulsion of teeth, Periodontal disease, After tumor resection), congenital alveolar defects, vertically deficient edentulous ridge in maxillary or mandibular anterior region with
* Allen Type A moderate vertical ridge deficiency (3-6mm)

Exclusion Criteria

* Medically compromised patients
* Subjects who underwent radiotherapy or chemotherapy
* Smokers and
* Radiographic presence of less than 5mm of anterior maxillary and mandibular bone height

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
height of the residual bone | From baseline to 6months.
  In radiographs, height of the residual bone will be taken as preoperative height. The gain in height of bone will be estimated after 6-months as postoperative bone height.

SECONDARY OUTCOMES:
Degree of inflammation in gingiva | From baseline to 2-months
  Degree of inflammation: degree of inflammation around the orthodontic implant was recorded by using the modified gingival index; 0 = normal gingiva; 1 = mild inflammation- slight change in color, slight edema, no bleeding on tissue manipulation. 2 = moderate inflammation- redness, edema and bleeding on tissue manipulation 3 = severe inflammation- marked redness and edema with ulceration and tendency for spontaneous bleeding.

CONTACTS AND LOCATIONS:
Locations (1):
- Svs Institute of Dental Science, Hyderabad, Telangana, India